CLINICAL TRIAL: NCT06192238
Title: A National Multicenter Study of Adrenal Venous Sampling for the Subtype Diagnosis of Primary Aldosteronism in China
Brief Title: China National Study of Adrenal Venous Sampling
Acronym: CNAVS
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xiongjing Jiang, professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 20231120
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Hyperaldosteronism
Keywords: Adrenal venous sampling; Hyperaldosteronism; Antecubital approach; Femoral approach; Pathological results
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adrenal Venous Sampling: Patients with Primary Aldosteronism (PA) undergoing Adrenal Venous Sampling via antecubital approach or femoral approach to discriminate PA forms with unilateral from bilateral excess aldosterone production.
  Interventions: Procedure: adrenal venous sampling

INTERVENTIONS:
Procedure: adrenal venous sampling — Patients with Primary Aldosteronism (PA) undergoing Adrenal Venous Sampling via antecubital approach or femoral approach to discriminate PA forms with unilateral from bilateral excess aldosterone production.

SUMMARY:
This multicenter study intends to combine retrospective analysis and prospective registry to evaluate the success rate and safety of adrenal venous sampling (AVS) via antecubital and femoral approach for patients with primary aldosteronism. The consistency of AVS with pathological results and clinical outcomes, the factors affecting the success of AVS, and the optimal population for AVS will be aslo analyzed in this study.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is one of the most common causes of secondary hypertension, and its most common subtypes are aldosterone-producing adenoma and idiopathic hyperaldosteronism, which account for 95% to 98% of PA. Subtype diagnosis is crucial for the treatment of primary aldosteronism, which conducts the appropriate treatment strategy. Currently, adrenal venous sampling (AVS) serves as the gold standard for subtyping of PA. How to improve the success rate of AVS has been a hot topic in the field of primary aldosteronism. This multicenter registry study intends to combine retrospective analysis and prospective registry to evaluate the success rate and safety of AVS via antecubital and femoral approach for patients with primary aldosteronism. The consistency of AVS with pathological results and clinical outcomes, the factors affecting the success of AVS, and the optimal population for AVS will be also analyzed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 65 with no limits in sex;
2. Patients with confirmed primary aldosteronism;
3. Patients or their legal representatives sign written informed consent approved by the ethics committee；

Exclusion Criteria:

1. Severe comorbidity, including stroke, myocardial infarction, heart failure, severe valvular heart disease, liver cirrhosis, and metastatic tumor within the previous 3 months；
2. An estimated glomerular filtration rate <45 ml/min/1.73 m2, or serum creatinine >176 μmol/L；
3. Patients who refuse adrenalectomy;
4. Suspected of having an adrenocortical carcinoma;
5. Allergy to contrast agent;
6. Pregnant, nursing, or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed primary aldosteronism aged from 18 to 65 with no limits in sex
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The success rate of bilateral adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)

SECONDARY OUTCOMES:
The success rate of left adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)
The success rate of right adrenal venous sampling | At AVS procedure
  Successful sampling will be defined by high selectivity index (cortisol in the adrenal vein/cortisol in inferior vena cava >2 without ACTH simulation)
Selection of intraoperative catheter | At AVS procedure
  Types of catheter at the time of Adrenal Venous Sampling via antecubital approach or femoral approach
Time of the procedure | At AVS procedure
  Time of the procedure
Time of fluoroscopy | At AVS procedure
  Time of fluoroscopy
The contrast agent dosage | At AVS procedure
  The contrast agent dosage
the incidence of complications | 1 week after AVS procedure
  Complications related to adrenal vein cannulations (adrenal vein hematoma, inferior vena cava dissection, puncture site hematoma, etc)
the cost of the procedure | At AVS procedure
  the cost of the procedure
pathological results（If the patient underwent adrenalectomy） | 1 week After AVS procedure
  Pathological types of primary aldosteronism（to compare the consistency between adrenal venous sampling results and histopathological results if the patients underwent adrenalectomy.）

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (48):
- China (48):
  - Chuiyangliu Hospital affiliated to Tsinghua University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - People's Hospital Affiliated to ChongqingThree Gorges Medical college, Chongqing, Chongqing Municipality
  - Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Forth People's Hosptal of Nanhai District of Foshan City, Foshan, Guangdong
  - Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Guangzhou, Guangdong
  - Shenzhen Third People's Hospital，Shenzhen, Guangdong Province 518112, China, Shenzhen, Guangdong
  - Shenzhen Dapeng New District Kuiyong People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Nanning Third People's Hospital, Nanning, Guangxi
  - The Second Affiliated Hospital Of Guizhou Medical University, Kaili, Guizhou
  - Tangshan hongci Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou Central Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou Yihe Hospital, Zhengzhou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Xiangyang Central Hospital, Affiliated Hospital of Hubei University of Arts and Science, Xiangyang, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Provincial People's Hospital (The First Affiliated Hospital of Nanchang Medical College), Nanchang, Jiangxi
  - Jilin Province FAW General ospital, Changchun, Jilin
  - Frist Aiffiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - Qinghai Province Cardiovascular and Cerebrovascular Disease Specialist Hospital, Xining, Qinghai
  - Xi'an People's Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - People's Hospital of Donga County, Shandong Province, Liaocheng, Shandong
  - Shanghai Institute of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Putuo District Central Hospital, Shanghai, Shanghai Municipality
  - The second hospital of Shanxi medical unversity, Taiyuan, Shanxi
  - The Affiliated Hospital of Southwest Jiaotong University, The Third People's Hospital of Chengdu, Chengdu, China, Chengdu, Sichuan
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital,, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality
  - Yili Kazak Autonomous Prefecture Friendship Hospital, Yili Kazak Autonomous Prefecture, Xinjiang
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan
  - Zhejiang Hospital, Hangzhou, Zhejiang